CLINICAL TRIAL: NCT02857426
Title: A Phase 2, Open-label, Single-arm, Two-cohort Study of Nivolumab in Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL) or Relapsed/Refractory Primary Testicular Lymphoma (PTL)
Brief Title: A Study of Nivolumab in Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL) and Relapsed/Refractory Primary Testicular Lymphoma (PTL)
Acronym: CheckMate 647
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-647; 2016-000894-19 (EudraCT Number)
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab for population with PCNSL (Experimental): Specified dose on specified days
  Interventions: Drug: Nivolumab
- Nivolumab for population with PTL (Experimental): Specified dose on specified days
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
  Other Names: BMS-936558; Opdivo

SUMMARY:
The purpose of this study is to determine whether Nivolumab is effective in the treatment of Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL) and Relapsed/Refractory Primary Testicular Lymphoma (PTL)

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Pathologically confirmed PCNSL or PTL who failed or did not respond to at least 1 line of systemic therapy
* Measurable disease requirements on scans:

PCNSL subjects should have at least one measurable extranodal brain lesion; PTL subjects should have at least 1 measurable extranodal lesion or nodal lesion

* Have tumor tissue for PD-L1 expression testing
* Must have a Karnofsky performance status of 70-100

Exclusion Criteria:

* a) Intraocular PCNSL without evidence of brain disease b) PCNSL patients who cannot undergo MRI assessments c) PCNSL patients with systemic disease
* Patients with certain diseases such as active autoimmune disease, type I diabetes, hypothyroidism that needs hormone replacement, active infection, psychiatric disorder
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

PCNSL, and PTL subjects with brain or spinal cord lesion who have received doses of more than 2 mg/day of dexamethasone or equivalent within the 14 days period prior to the first dose of nivolumab are excluded

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (50):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City Of Hope Medical Center, Duarte, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center & Research Inst, Inc, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
- Brazil (3):
  - Instituto Do Cancer Mae De Deus / Cor Hospital Mae De Deus, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio Xii Hosp Cancer De Barretos, Barretos, São Paulo
  - Hospital Das Clinicas - Fmusp, São Paulo
- Canada (3):
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHU de Quebec, Québec, Quebec
- I. interni klinika - klinika hematologie 1. LF UK a VFN v Praze, Prague, Czechia
- France (9):
  - Local Institution, Bordeaux
  - Local Institution, Caen
  - Local Institution, La Tronche
  - Local Institution, Lille
  - Local Institution, Paris
  - Centre Hospitalier Lyon Sud - UPCO, Pierre-Bénite
  - Local Institution, Rennes
  - Local Institution, Saint-Cloud
  - Local Institution, Tours
- Klinikum Stuttgart, Stuttgart, Germany
- Local Institution, Hong Kong, Hong Kong
- Hungary (3):
  - Local Institution, Budapest
  - Belgyogyaszati Onkologia OOI, Budapest
  - Local Institution, Debrecen
- Israel (4):
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Petah Tikva
  - Local Institution, Tel Aviv
- Italy (3):
  - Irccs Ospedale S. Raffaele, Milan
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano (milano)
- Japan (7):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Hidaka-shi, Saitama
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Kotoku, Tokyo
  - Local Institution, Mitaka-shi, Tokyo
  - Local Institution, Yamagata
- Local Institution, Moscow, Russia
- Local Institution, Singapore, Singapore

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 PCNSL participants treated.
  19 PTL participants treated.
Groups:
- PCNSL Cohort: Nivolumab dosed to participants with relapsed/refractory Primary Central Nervous System Lymphoma (PCNSL).
  Nivolumab 240 mg was given every 2 weeks for 8 cycles. Beginning with Cycle 9, nivolumab 480 mg was given every 4 weeks for a total therapy duration of 2 years, or until progressive disease, unacceptable toxicity, or withdrawal of consent. Nivolumab was administered as a 30-minute infusion.
- PTL Cohort: Nivolumab dosed to participants with relapsed/refractory Primary Testicular Lymphoma (PTL).
  Nivolumab 240 mg was given every 2 weeks for 8 cycles. Beginning with Cycle 9, nivolumab 480 mg was given every 4 weeks for a total therapy duration of 2 years, or until progressive disease, unacceptable toxicity, or withdrawal of consent. Nivolumab was administered as a 30-minute infusion.
Period: Overall Study
Arm/Group | PCNSL Cohort | PTL Cohort
Started (Started = received treatment) | 47 | 19
Completed (Completed = continuing in the treatment period) | 0 | 0
Not Completed | 47 | 19
Not completed — Disease progression | 34 | 13
Not completed — Study drug toxicity | 4 | 1
Not completed — Death | 1 | 0
Not completed — Adverse event unrelated to study drug | 6 | 2
Not completed — Participant withdrew consent | 1 | 1
Not completed — Maximum clinical benefit | 1 | 0
Not completed — Completed treatment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCNSL Cohort | PTL Cohort | Total
Number analyzed (Participants) | 47 | 19 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (10.1) | 66.7 (8.6) | 66.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 0 | 20
  Male | 27 | 19 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 33 | 11 | 44
  Unknown or Not Reported | 13 | 8 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 37 | 12 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: BICR-Assessed Objective Response Rate (ORR)
Description: Percentage of participants with a confirmed objective response rate (ORR) by blinded independent central review (BICR) assessment was analyzed and reported for both PCNSL and PTL patient populations.
  This endpoint is further defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR), based on the IPCG Criteria for PCNSL and Lugano 2014 response evaluation for PTL, divided by the number of treated participants within each cohort.
Time Frame: Up to approximately 51 months
Population: All treated PCNSL and PTL participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PCNSL Cohort | PTL Cohort
Number analyzed (Participants) | 47 | 19
Percentage of participants | 6.4 [1.3 to 17.5] | 26.3 [9.1 to 51.2]

2. Secondary Outcome: BICR-Assessed Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from first dosing date to the date of the first documented progression using the IPCG Criteria for PCNSL and Lugano 2014 response evaluation for PTL, as determined by BICR, or death due to any cause, whichever occurs first.
Time Frame: Up to approximately 51 months
Population: All treated PCNSL and PTL participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PCNSL Cohort | PTL Cohort
Number analyzed (Participants) | 47 | 19
Months | 1.41 [1.08 to 1.74] | 1.72 [1.15 to 6.28]

3. Secondary Outcome: Investigator-Assessed Objective Response Rate (ORR)
Description: Percentage of participants with a confirmed objective response rate (ORR) by investigator assessment was analyzed and reported for both PCNSL and PTL patient populations.
  This endpoint is further defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR), based on the IPCG Criteria for PCNSL and Lugano 2014 response evaluation for PTL, divided by the number of treated participants within each cohort.
Time Frame: Up to approximately 51 months
Population: All treated PCNSL and PTL participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PCNSL Cohort | PTL Cohort
Number analyzed (Participants) | 47 | 19
Percentage of participants | 10.6 [3.5 to 23.1] | 26.3 [9.1 to 51.2]

4. Secondary Outcome: Investigator-Assessed Duration of Response (DOR)
Description: Duration of response (DOR) by investigator assessment was analyzed and reported for both PCNSL and PTL patient populations.
  This endpoint is further defined as the time from first response (CR or PR) to the date of initial objectively documented progression as determined using the IPCG Criteria for PCNSL and Lugano 2014 response evaluation for PTL, as determined by BICR, or death due to any cause, whichever occurs first.
Time Frame: Up to approximately 51 months
Population: All responders PCNSL and PTL participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PCNSL Cohort | PTL Cohort
Number analyzed (Participants) | 5 | 5
Months | 1.71 [0.72 to 7.10] | 20.63 [0.03 to NA] — only 3 DOR event observed

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was analyzed and reported for both PCNSL and PTL patient populations.
  OS is defined as the time from first dosing date to the date of death. For participants without documentation of death, OS will be censored on the last date the participant was known to be alive.
Time Frame: Up to approximately 51 months
Population: All treated PCNSL and PTL participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PCNSL Cohort | PTL Cohort
Number analyzed (Participants) | 47 | 19
Months | 6.77 [3.68 to 11.99] | 11.17 [2.60 to 24.41]

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose (up to approximately 48 months)
Groups:
- PCNSL Cohort Nivolumab 240 mg (Q2W): Nivolumab dosed to participants with relapsed/refractory Primary Central Nervous System Lymphoma (PCNSL).
  Nivolumab 240 mg was given every 2 weeks for 8 cycles. Beginning with Cycle 9, nivolumab 480 mg was given every 4 weeks for a total therapy duration of 2 years, or until progressive disease, unacceptable toxicity, or withdrawal of consent. Nivolumab was administered as a 30-minute infusion.
- PTL Cohort Nivolumab 240 mg (Q2W): Nivolumab dosed to participants with relapsed/refractory Primary Testicular Lymphoma (PTL).
  Nivolumab 240 mg was given every 2 weeks for 8 cycles. Beginning with Cycle 9, nivolumab 480 mg was given every 4 weeks for a total therapy duration of 2 years, or until progressive disease, unacceptable toxicity, or withdrawal of consent. Nivolumab was administered as a 30-minute infusion.
Arm/Group | PCNSL Cohort Nivolumab 240 mg (Q2W) | PTL Cohort Nivolumab 240 mg (Q2W)
All-Cause Mortality (participants affected / at risk) | 32/47 | 13/19
Serious Adverse Events (participants affected / at risk) | 33/47 | 15/19
Other Adverse Events (participants affected / at risk) | 40/47 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCNSL Cohort Nivolumab 240 mg (Q2W) (N=47) | PTL Cohort Nivolumab 240 mg (Q2W) (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 8
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 2 | 0
Hemianopia homonymous (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 2 | 0
Optic neuritis (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 4 | 1
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCNSL Cohort Nivolumab 240 mg (Q2W) (N=47) | PTL Cohort Nivolumab 240 mg (Q2W) (N=19)
Anaemia (Blood and lymphatic system disorders) | 13 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Bradycardia (Cardiac disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 1 | 1
Glaucoma (Eye disorders) | 0 | 2
Pupils unequal (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 7 | 0
Asthenia (General disorders) | 2 | 2
Fatigue (General disorders) | 12 | 2
Gait disturbance (General disorders) | 6 | 1
Mucosal inflammation (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 3 | 2
Pyrexia (General disorders) | 9 | 5
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 5 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 9 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Recall phenomenon (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 10 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 1
Blood creatinine increased (Investigations) | 3 | 1
Human rhinovirus test positive (Investigations) | 0 | 1
Lipase increased (Investigations) | 3 | 1
Lymphocyte count decreased (Investigations) | 6 | 0
Neutrophil count decreased (Investigations) | 5 | 1
Platelet count decreased (Investigations) | 5 | 1
Weight decreased (Investigations) | 4 | 0
White blood cell count decreased (Investigations) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Aphasia (Nervous system disorders) | 5 | 0
Ataxia (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 12 | 1
Hemiparesis (Nervous system disorders) | 5 | 0
Paraesthesia (Nervous system disorders) | 3 | 0
Seizure (Nervous system disorders) | 6 | 0
Somnolence (Nervous system disorders) | 3 | 0
Agitation (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 4 | 0
Confusional state (Psychiatric disorders) | 4 | 1
Depression (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 5 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 5 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Testicular swelling (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT02857426/Prot_001.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT02857426/SAP_000.pdf